CLINICAL TRIAL: NCT04774536
Title: Transplantation of CRISPRCas9 Corrected Hematopoietic Stem Cells (CRISPR_SCD001) in Patients with Severe Sickle Cell Disease
Brief Title: Transplantation of Clustered Regularly Interspaced Short Palindromic Repeats Modified Hematopoietic Progenitor Stem Cells (CRISPR_SCD001) in Patients with Severe Sickle Cell Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mark Walters, MD (Other)
Collaborators: University of California, Los Angeles (Other); University of California, Berkeley (Other)
Responsible Party: Sponsor-Investigator, Mark Walters, MD, Professor in Residence, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-33287
Record Dates: First submitted 2021-02-17; First posted 2021-03-01 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CRISPR_SCD001 Drug Product (Experimental): CRISPR_SCD001 Drug Product (autologous CD34+ cell-enriched population that contains cells modified by the CRISPR-Cas9 ribonucleoprotein) dose will be ≥3.0×106 CD34+ cells/kg recipient weight for each subject and the upper limit cell dose is 20 ×106 CD34+ cells/kg.
  Interventions: Drug: CRISPR_SCD001

INTERVENTIONS:
Drug: CRISPR_SCD001 — CRISPR_SCD001 is administered by IV infusion following myeloablative conditioning with busulfan.

SUMMARY:
This is an open label, non-randomized, 2-center, phase 1/2 trial of a single infusion of sickle allele modified cluster of differentiation (CD34+) hematopoietic stem progenitor cells (HSPCs) in subjects with in subjects ≥12 years old to 35 years old severe Sickle Cell Disease (SCD). The study will evaluate the hematopoietic stem cell transplantation (HSCT) using CRISPR/Cas9 edited red blood cells (known as CRISPR_SCD001 Drug Product).

DETAILED DESCRIPTION:
This is an open label, non-randomized, 2-center, phase 1/2 trial of a single infusion of sickle allele modified CD34+ HSPCs in subjects with severe SCD. The primary endpoint of the trial will determine the safety of CRISPR_SCD001 through a 3+3 design with staggered enrollment and a pause in enrollment for safety review after each of the first 3 patients has had drug product infused. After safety is assessed in the 3rd patient, enrollment of the next 3 patients will not be staggered. The first six subjects will be adults. If CRISPR_SCD001 is determined to be safe in the first six subjects, the trial will continue to enroll 3 adolescents 12 - 18 years of age to evaluate the safety in younger patients. The younger age cohort also will follow staggered enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 12.00 - 34.99 years of age (at time of consent) who have one or more of the following:

   1. History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea);
   2. History of at least 4 severe vaso-occlusive pain events in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea); painful episodes related to or any sickle-related acute event are acceptable; a severe painful vaso-occlusive event is defined as receiving analgesic treatment (opioid or other analgesic) for longer than 24 -hours in a hospital or emergency room (ER) observation unit visit or at least 2 visits in a day unit or ER over 72 hours with both visits requiring intravenous analgesics.
2. Participants must have adequate physical function as measured by all of the following:

   1. Karnofsky performance score ≥60.
   2. Cardiac function: Left ventricular ejection fraction (LVEF) >40%; or LV shortening fraction > 26% by cardiac echocardiogram or by (multiple-gated acquisition) MUGA scan.
   3. Pulmonary function: Pulse oximetry with a baseline O2 saturation of ≥85% and diffusion capacity of lung for carbon monoxide(DLCO) > 40% (corrected for hemoglobin).
   4. Renal function: Serum creatinine ≤ 1.5 x upper limit of normal for age and estimated or measured creatinine clearance ≥ 70 mL/min/1.73 m2.
   5. Hepatic function:

   i. Serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory. Participants with hyperbilirubinemia as the result of hyperhemolysis, or a severe drop in hemoglobin post blood transfusion, are not excluded.

   ii. Alanine aminotransferase (ALT) and aspartate aminotransferase (AS < 5 times upper limit of normal as per local laboratory.

   f. Liver MRI using a validated methodology per institutional preference (T2* or R2* or by ferriscan [R2 MRI]) for estimation of hepatic iron content is required for participants who are currently receiving ≥8 packed red blood cell transfusions per year for ≥1 year or have received ≥20 packed red blood cell transfusions (lifetime cumulative). Participants who have hepatic iron content ≥ 8 mg Fe/g liver dry weight by liver MRI must have a Gastroenterology/hepatology consultation with liver biopsy and histological examination including documentation of the absence of cirrhosis, bridging fibrosis[1], and active hepatitis.
3. Written informed consent or assent obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Participants with uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
2. Participants with evidence of HIV infection or seropositivity for HIV or active hepatitis B or C.
3. Participants who have received a Hematopoietic Cell Transplant (HCT)
4. Participants who have received a solid organ transplant.
5. Participants who have participated in another clinical trial in which the participant received an investigational or off-label use of a drug or device within 3 months prior to enrollment.
6. Females who are pregnant or breast feeding.
7. Females of child bearing potential (to include all female participants > 10 years of age, unless postmenopausal for a minimum of 1 year before the time of consent or surgically sterilized) who do not agree to practice two (2) effective methods of contraception at the same time, or who do not agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject, from the time of signing of informed consent through 12 months post-stem cell infusion.
8. Males (even if surgically sterilized) who do not agree to practice effective barrier contraception, or who do not agree to practice true abstinence from the time of signing informed consent through 12 months post-stem cell infusion.
9. Participants who have had a stroke OR who are receiving red blood cell (RBC) transfusions to prevent primary stroke or silent cerebral infarction.
10. Patients who have a human leukocyte antigen identical (HLA-ID) sibling donor
11. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
12. Any non-homozygous sickle hemoglobin (HbSS) genotype of SCD

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events and grade 3 or higher serious adverse events, using the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) | 24 months post-transplant
  The adverse event rate will be summarized using descriptive statistics, together with 95% confidence intervals where appropriate. No formal statistical hypothesis testing will be performed. Adverse events defined: failure of engraftment, malignant clonal expansion related to genomic editing or death.

SECONDARY OUTCOMES:
Change in the annualized vaso-occlusive pain event (VOE) rates. | 24 months pre-transplant to 24 months post-transplant
  Change in the annualized vast-occlusive pain event (VOE) rates comparing the 24 months before with 24 months after the infusion of drug product.
Graft rejection defined as having an absolute neutrophil count (ANC) < 500 at 42 days post-infusion | 42 days post-transplant
  A delay in platelet and/or neutrophil engraftment will be captured.
Time to neutrophil recovery defined as the first of 3 measurements on different days when the patient has an absolute neutrophil count (ANC) of ≥500/µL after transplant. | 24 months post-transplant
  Neutrophil recovery as part of the overall hematological recovery.
Time to platelet recovery is defined as the first day of a minimum of 3 measurements on different days that the patient has achieved a platelet count > 50,000/µL AND did not receive a platelet transfusion in the previous 7 days. | baseline, through 24 months post-transplant
  Platelet recovery as part of the overall hematological recovery.
Rate of improvement in Hemoglobin S (HbS) fraction as measured by hemoglobin electrophoresis, as percent of total. | baseline, through 24 months post-transplant
  Hemolysis markers.
Rate of normalization in hemoglobin (hgb) level as measured by clinical hematology (laboratory) test. | baseline, through 24 months post-transplant
  Hemolysis markers.
Rate of normalization of lactate dehydrogenase (LDH), reticulocyte count, and haptoglobin, as measured by clinical hematology and serum chemistry (laboratory) tests. | baseline, through 24 months post-transplant
  Hemolysis markers.
Frequency of hepatic veno-occlusive disease (VOD) as measured by Seattle or Baltimore Criteria for VOD Diagnosis. | 24 months post-transplant
  Hematologic and non-hematologic toxicities of autologous transplantation with CRISPR-Cas9 sickle-corrected HSPCs.
Frequency of hepatic idiopathic pneumonia syndrome (IPS) as measured by the Idiopathic pneumonia syndrome (IPS) criteria. | 24 months post-transplant
  Hematologic and non-hematologic toxicities of autologous transplantation with CRISPR-Cas9 sickle-corrected HSPCs.
Frequency of central nervous system (CNS) toxicity (reversible posterior leukoencephalopathy syndrome [RPLS] or posterior reversible encephalopathy syndrome [PRES], hemorrhage, and seizures). | 24 months post-transplant
  Hematologic and non-hematologic toxicities of autologous transplantation with CRISPR-Cas9 sickle-corrected HSPCs.
Frequency of cytomegalovirus (CMV) infection, invasive fungal infection, and any other serious viral or bacterial infection | 24 months post-transplant
  Hematologic and non-hematologic toxicities of autologous transplantation with CRISPR-Cas9 sickle-corrected HSPCs.
Frequency of sickle gene-editing (correction and insertion/deletion) and off-target site-1 editing in marrow and peripheral blood mononuclear cells. | 3 months, 1 and 2 years post-transplant
  Stability of gene-editing in hematopoietic cells by genotyping studies.

OTHER OUTCOMES:
Rate of sickle-related events other than severe VOE and end organ function. | 24 months post-infusion
  Rate of sickle-related complications after infusion
Patient-reported quality of life (pain and fatigue domains) as measured by the use of Patient Reported Outcome Measurement Information System (PROMIS) modules. | baseline, and 1 and 2 years post-transplant
  Change in quality of life score at baseline (prior to the initiation of hydroxyurea), 1 year and 2 years post-stem cell infusion accessed using Patient Reported Outcome Measurement Information System (PROMIS) modules. The PROMIS modules rate the following areas:
  * Physical Function and Sleep Quality on a scale of 1 (not good) to 5 (good).
  * Anxiety, Depression, Fatigue, Pain Interference and the Ability to Participate in Social Roles and Activities on a scale of 1 (never) to 5 (always).
  * Pain Intensity on a scale from 0 (no pain) to 10 (worst pain imaginable).
Change from baseline in cardiac-pulmonary function via pulmonary function tests | Through 1 and 2 years post-transplant
Change from baseline in cardiac-pulmonary function via echocardiogram (tricuspid regurgitant jet velocity [TRJV], LVEF). | Through 1 and 2 years post-transplant
Change from baseline in meters walked during 6-minute walk test (6MWD) | Through 1 and 2 years post-transplant
Event-free survival defined as survival without clinical and hematological evidence of the underlying Sickle Cell Disease (SCD) | 1 and 2 years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Mark Walters, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital, Oakland, California

IPD SHARING:
Plan to Share IPD: No